CLINICAL TRIAL: NCT03448848
Title: Role of Branched-chain Amino Acids Infusion as Adjunct Therapy Post Liver Surgery for Patients in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, ICU, Consultant of Intensive care medicine, Ph D, National Hepatology & Tropical Medicine Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BCAA
Record Dates: First submitted 2018-01-02; First posted 2018-02-28 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Liver Function Post BCAA Infusion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Experimental)
  Interventions: Drug: BCAA preparation Intravenous infusion
- control (Placebo Comparator)
  Interventions: Drug: sterile normal saline

INTERVENTIONS:
Drug: BCAA preparation Intravenous infusion — BCAA IVi in a dose 0.5-1 gm/Kg/day for 2-5 days post liver surgery versus sterile normal saline in a volume equal to the study drug
  Arms: study
Drug: sterile normal saline — sterile normal saline in a volume equal to the study drug
  Arms: control

SUMMARY:
The purpose of this study is to evaluate the impact of intravenous BCAAs infusion as adjunct therapy post liver surgery in intensive care unit (ICU).

DETAILED DESCRIPTION:
Patients will be enrolled in the study&randomly assigned in a 1:1 manner to receive either intravenous (IV) BCAAs in a dose of 0.5-1gm/Kg/day for at least 48hours up to maximum 5 days immediately post-operative or placebo (sterile normal saline in a volume equal to the study drug).

All demographic data will be obtained including the patients' age, sex, weight,associated co-morbidities (diabetes mellitus & hypertension), the presence of chronic liver disease (CLD), Child-Pugh score, Sequential Organ Failure Assessment (SOFA), the type of liver surgery, & nutritional status according to nutritional risk screening 2002 (NRS 2002); well-nourished if NRS 2002 < 3 while malnourished if NRS 2002 ≥ 3 prior BCAAs infusion.

Vital signs including the heart rate, mean arterial pressure (MAP), central venous pressure (CVP), arterial oxygen saturation (SaO2), insulin requirements, urine volume & fluid balance will be recorded on admission (day 0), then will be followed up and recorded at regular intervals during treatment on 1, 3, 5 &7days.

Laboratory investigations including the complete blood profile (white blood cells, band%, lymphocytes), prothrombin time (PT), liver enzymes; Aspartate aminotransferase (AST), Alanine aminotransferase (ALT),serum bilirubin, serum albumin, C-reactive protein (CRP)& kidney functions will be recorded at randomization as a baseline (day 0)& will be assessed on day 0,1, 3, 5 & 7 of the study. Thirty-day survival & infectious morbidity will be followed by phone calls to the patient or one of his/her first-degree relatives.

ELIGIBILITY:
Inclusion Criteria:

* The subjects are adults aged between 18& 75years who are admitted to the ICU of National Hepatology & Tropical Medicine Research Institute (NHTMRI) post liver surgery e.g. hepatocellular carcinoma, liver hemangioma, hydatid resection, segmentectomy, partial hepatectomy as in donor for living donated liver transplant.

Exclusion Criteria:

* if pregnant.
* hemodynamic instability requiring circulatory support.
* need for dose of BCAAs > 1gm/Kg/day or < 0.5 gm/Kg/day.
* severe malnutrition; body mass index (BMI < 16).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
effect on liver function tests | within one week post liver surgery
  improvement of liver function tests, AsT
effect on liver function tests | within one week post liver surgery
  improvement of ALT
effect on liver function tests | within one week post surgery
  Improvement of total bilirubin
effect on liver function tests | within one week post surgery
  improvement of alkaline phosphatase
effect on liver function tests | within one week post surgery
  improvement of prothrombin time
Child-Pugh score post-surgery. | within one week post surgery
  Improvement with BCAA infusion
SOFA score post-surgery | within one week post surgery
  improvement with BCAA infusion

SECONDARY OUTCOMES:
30-day infectious morbidity Infectious morbidity | 30 days post surgery
  occurrence of infections post surgery
non infectious morbidity | 30 days
  occurrence of hepatic encephalopathy, ruptured esophageal varices, ascites requiring diuretic agent for control, wound dehiscence, intra-abdominal bleeding, intestinal obstruction, renal failure, pleural effusion, need mechanical ventilation, blood sugar control & nutritional status change.
ICU stay. length of ICU stay, length of hospital stay & 28day mortality. length of ICU stay, length of hospital stay & 28day mortality. length of ICU stay, length of hospital stay & 28day mortality. | within two weeks post surgery
  Length of ICU stay in days
Hospital stay. length of ICU stay, length of hospital stay & 28day mortality. length of ICU stay, length of hospital stay & 28day mortality. length of ICU stay, length of hospital stay & 28day mortality. | within two weeks post surgery
  Length of hospital stay in days
mortality | 28 day
  28-day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- NHTMRI, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mahmoud EIE, Awdallah FF. Prospective randomized, placebo-controlled study: role of branched-chain amino acids infusion as adjunct therapy post-liver surgery for patients in the intensive care unit. BMC Gastroenterol. 2025 Jun 19;25(1):439. doi: 10.1186/s12876-025-03696-3. PMID 40537743